CLINICAL TRIAL: NCT02531139
Title: The Effect of Blood Pressure on Cerebral Perfusion and Oxygenation During Vascular Surgery
Brief Title: The Effect of Blood Pressure on Cerebral Perfusion During Vascular Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not feasible.
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Niels Damkjær Olesen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NDOlesen
Record Dates: First submitted 2015-08-14; First posted 2015-08-24 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Anesthesia; Peripheral Arterial Diseases
Keywords: Cerebrovascular Circulation; Anesthesia; Blood pressure; Peripheral Arterial Diseases
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAP maintained at 80 mmHg (Experimental): During anesthesia MAP is maintained at 80 - 90 mmHg MAP using continuous infusion of phenylephrine.
  Interventions: Other: MAP maintained at 80 mmHg
- MAP maintained at 60 mmHg (Active Comparator): During anesthesia MAP is maintained at minimum of 60 mmHg using continuous infusion of phenylephrine.
  Interventions: Other: MAP maintained at 60 mmHg

INTERVENTIONS:
Other: MAP maintained at 80 mmHg — Intervention group, MAP is maintained at 80 - 90 mmHg during anesthesia using continuous infusion of phenylephrine.
  Arms: MAP maintained at 80 mmHg
Other: MAP maintained at 60 mmHg — Control group, MAP is maintained at minimum of 60 mmHg during anesthesia using continuous infusion of phenylephrine.
  Arms: MAP maintained at 60 mmHg

SUMMARY:
Anesthesia reduces blood pressure and cerebral blood flow is normally considered to be maintained despite marked changes in blood pressure. Vascular surgical patients are often elderly, have high blood pressure and atherosclerosis and in these patients cerebral blood flow may decrease if blood pressure is reduced during anesthesia. The purpose of this study is to assess the effect of blood pressure for preservation of cerebral blood flow during anesthesia in vascular surgery. The hypothesis is that in vascular surgical patients, during anesthesia, cerebral blood flow is higher with blood pressure maintained at a higher level than that used in normal clinical practice.

DETAILED DESCRIPTION:
Background: Induction of anesthesia reduces mean arterial pressure (MAP) and cerebral blood flow is normally considered to be maintained by cerebral autoregulation despite changes in MAP between 60 - 150 mmHg and standard of care during anesthesia is to maintain MAP above 60 mmHg. Vascular surgical patients are often elderly with hypertension and atherosclerotic manifestations that may impair cerebral autoregulation of importance for anesthesia-induced reduction in blood pressure.

Objective: To assess the effect of MAP for preservation of cerebral blood flow and oxygenation during vascular surgery.

Hypothesis: The primary hypothesis is that during general anesthesia in vascular surgical patients, cerebral blood flow velocity and oxygenation is higher with MAP maintained at 80-90 mmHg, compared with a MAP maintained at a minimum of 60 mmHg.

MAP is controlled in both groups using continuous infusion of phenylephrine. Phenylephrine is used as a tool in order to assess the effect of MAP on the cerebral circulation. In both groups, central blood volume is optimized by infusion of lactated Ringer´s solution using a goal directed fluid therapy following induction of anaesthesia and before commencement of phenylephrine infusion.

Trial size: The investigators will include 40 participants (2 x 20) in order to detect or reject a 20% difference in middle cerebral artery velocity with a type I error risk of 5% and a type II error risk of 20% (power at 80%). Interim analysis will be conducted after inclusion of 20 patients (2 x 10). Excluded patients will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing one of the following vascular surgical interventions in general anesthesia: Infra-inguinal bypass, femoro-femoral cross-over bypass or iliofemoral bypass surgery.
* Age > 18 years. Informed consent

Exclusion Criteria:

* Use of monoamine oxidase inhibitors
* Allergy to phenylephrine
* Patients that cannot cooperate during examination
* Dementia defined as Mini-Mental State Examination < 24
* Anesthesia within the last 30 days
* Alcohol consumption at or above 420 grams per week
* Lack of fluency in written and spoken Danish
* Severe hearing and vision impairment
* Neurological disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Middle cerebral artery blood velocity | During surgery
  Middle cerebral artery blood velocity measured in [cm/s] assessed by transcranial Doppler. Changes in middle cerebral artery blood velocity reflects changes in cerebral blood flow.

SECONDARY OUTCOMES:
Change in serum S100B as compared between subjects in the control- and intervention groups | Blood is sampled 10 min prior to induction of anesthesia and at the end of surgery
  Serum concentrations of S100B, a marker of neuronal injury
Change in serum neuron-specific enolase as compared between subjects in the control- and intervention groups | Blood is sampled 10 min prior to induction of anesthesia and at the end of surgery
  Serum concentrations of neuron-specific enolase, a marker of neuronal injury
Regional cerebral oxygenation as compared between subjects in the control- and intervention groups | During surgery
  Frontal lobe oxygenation measured as the percentage of oxyhemoglobin of total hemoglobin [%] evaluated by near-infrared spectroscopy
Cardiac output as compared between subjects in the control- and intervention groups | During surgery
  Cardiac output measured in [l/min] evaluated by pulse contour analysis of the arterial blood pressure curve
Stroke volume as compared between subjects in the control- and intervention groups | During surgery
  Stroke volume measured in [ml/min] evaluated by pulse contour analysis of the arterial blood pressure curve

CONTACTS AND LOCATIONS:
Overall Officials: Niels D. Olesen, MD, Principal Investigator — Rigshospitalet, Anæstesi og Operationsklinikken 2043, Denmark
Locations (1):
- Rigshospitalet, Anæstesi og Operationsklinikken 2043, Copenhagen Ø, Denmark